CLINICAL TRIAL: NCT01751165
Title: Open-label Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults Aged 50 Years or Older
Brief Title: Safety and Immunogenicity of Different Dosing Schedules of GlaxoSmithkline (GSK) Biologicals' Herpes Zoster (HZ) Vaccine in Adults 50 Years of Age or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116697; 2012-004456-11 (EudraCT Number)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-06

CONDITIONS: Herpes Zoster
Keywords: ≥ 50 years of age; Herpes zoster; Safety; Immunogenicity; Adults
MeSH Terms: conditions — Herpes Zoster

ARMS (3):
- HZ/su-0,2 Group (Experimental): Subjects will receive HZ/su vaccine on a 0,2-month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- HZ/su-0,6 Group (Experimental): Subjects will receive HZ/su vaccine on a 0,6-month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- HZ/su-0,12 Group (Experimental): Subjects will receive HZ/su vaccine on a 0,12-month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A

INTERVENTIONS:
Biological: Herpes zoster vaccine GSK1437173A — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of the GSK Biologicals' HZ vaccine 1437173A administered on either a 0,2-; 0,6- or 0,12-month schedule in adults aged 50 years or above, as the immunogenicity of the HZ vaccine administered at intervals longer than two months is not known.

DETAILED DESCRIPTION:
Subjects in each group will be stratified by age with a minimum of 35 subjects in each stratum (50-59 years of age (YOA) stratum, 60-69 YOA stratum and ≥ 70 YOA stratum).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female aged 50 years or older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, a prednisone dose of < 20 mg/day, or equivalent, is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a live vaccine in the period starting 30 days before and ending 30 days after either dose of study vaccine.
* Administration or planned administration of a non-replicating vaccine within eight days prior to or within 14 days after either dose of study vaccine.
* Administration of long-acting immune-modifying drugs (e.g. infliximab) within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Previous vaccination against varicella or HZ (either registered product or participation in a previous vaccine study).
* Planned administration during the study of an HZ or varicella vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* History of HZ.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g. malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g. medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C (99.5°F) for oral, axillary or tympanic route, or ≥ 38.0°C (100.4°F) for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Significant underlying illness that, in the opinion of the investigator, would be expected to prevent completion of the study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Pregnant or lactating female.
* Female planning to become pregnant during the entire treatment period and for two months after completion of the vaccination series, or planning to discontinue contraceptive precautions (if of childbearing potential).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-03-12; Primary Completion 2014-05-22 (Actual); Study Completion 2015-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (3):
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Uniontown, Pennsylvania
- GSK Investigational Site, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lal H, Poder A, Campora L, Geeraerts B, Oostvogels L, Vanden Abeele C, Heineman TC. Immunogenicity, reactogenicity and safety of 2 doses of an adjuvanted herpes zoster subunit vaccine administered 2, 6 or 12 months apart in older adults: Results of a phase III, randomized, open-label, multicenter study. Vaccine. 2018 Jan 2;36(1):148-154. doi: 10.1016/j.vaccine.2017.11.019. Epub 2017 Nov 22. PMID 29174683
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK1437173A-0,2 M Group: Healthy subjects aged 50 or older received the GSK1437173A vaccine administered intramuscularly on a 0,2-month schedule.
- GSK1437173A-0,6 M Group: Healthy subjects aged 50 or older received the GSK1437173A vaccine administered intramuscularly on a 0,6-month schedule.
- GSK1437173A-0,12 M Group: Healthy subjects aged 50 or older received the GSK1437173A vaccine administered intramuscularly on a 0,12-month schedule.
Period: Overall Study
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Started | 119 | 119 | 116
Completed | 117 | 116 | 113
Not Completed | 2 | 3 | 3
Not completed — Adverse event, serious fatal | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Serious adverse event | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group | Total
Number analyzed (Participants) | 119 | 119 | 116 | 354
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.9) | 64 (8.6) | 64.1 (9.2) | 64.2 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 77 | 79 | 246
  Male | 29 | 42 | 37 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to Anti-glycoprotein E (Anti-gE) Antibodies as Determined by the Enzyme-linked Immunosorbent Assay (ELISA).
Description: Vaccine response was defined as: for initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL); for initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
  The objective required a comparison of VRR between 0,6-months and 0,12-months schedules.
Time Frame: At one month (M1) after Dose 2
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all subjects who had met all eligibility criteria and for whom data concerning immunogenicity outcome measures were available.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 114 | 110
Subjects | 110 | 104

2. Primary Outcome: Concentrations of Antibodies Against Anti-gE as Determined by ELISA.
Time Frame: At one month (M1) after Dose 2
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity, which included all evaluable subjects for whom the pre vaccination and one month post dose 2 time point data were obtained from ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 118 | 114 | 111
mIU/mL | 44376.3 [39697 to 49607.2] | 38153.7 [34205.8 to 42557.3] | 37435.8 [30813.8 to 45480.8]
Statistical Analysis 1: Comparison: GSK1437173A-0,2 M Group vs GSK1437173A-0,6 M Group; To demonstrate the non-inferiority in terms of anti-gE humoral immune response one month post-dose 2 given according to a 0,6-month schedule compared to a 0,2-month schedule; Test type: Non-Inferiority or Equivalence — Non-nferiority criteria: The upper limit (UL) of the 97.5% confidence interval (CI) for the anti-gE ELISA geometric mean concentration (GMC) ratio (0,2-month schedule over 0,6-month schedule) at one month post-dose 2 had to be below 1.5; ANCOVA; Adjusted GMC ratio = 1.16, 97.5% CI 2-sided [0.98 to 1.39]
Statistical Analysis 2: Comparison: GSK1437173A-0,2 M Group vs GSK1437173A-0,12 M Group; To demonstrate the non-inferiority in terms of anti-gE humoral immune response one month post-dose 2 given according to a 0,12-month schedule compared to a 0,2-month schedule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.19, 97.5% CI 2-sided [0.93 to 1.53]

3. Secondary Outcome: Concentrations of Antibodies Against Anti-gE as Determined by ELISA.
Time Frame: Prior (PRE) to vaccination and twelve (M12) post Dose 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 118 | 115 | 110
mIU/mL
  Anti-gE, PRE [N=118,114,110] | 1079.1 [891.9 to 1305.5] | 1066.1 [891.3 to 1275.3] | 1019.4 [858.6 to 1210.2]
  Anti-gE, M12 [N=117,115,110] | 14245.4 [12450.8 to 16298.6] | 12911.5 [11412.7 to 14607.2] | 11892.1 [10236.4 to 13815.6]

4. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Solicited local symptoms assessed include pain, redness and swelling. "Grade 3 pain" was defined as crying when limb was moved/spontaneously painful. "Grade 3 swelling/redness" was defined as swelling/redness larger than (>) 100 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 7 day period (Days 0-6) following each dose (D)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects
  Any Pain, D1 [N=119,119,115] | 84 | 77 | 80
  Grade 3 Pain, D1 [N=119,119,115] | 1 | 0 | 2
  Any Redness, D1 [N=119,119,115] | 37 | 39 | 32
  Grade 3 Redness, D1 [N=119,119,115] | 0 | 0 | 1
  Any Swelling, D1 [N=119,119,115] | 17 | 23 | 25
  Grade 3 Swelling, D1 [N=119,119,115] | 0 | 0 | 0
  Any Pain, D2 [N=118,117,111] | 71 | 83 | 87
  Grade 3 Pain, D2 [N=118,117,111] | 6 | 6 | 10
  Any Redness, D2 [N=118,117,111] | 28 | 27 | 37
  Grade 3 Redness, D2 [N=118,117,111] | 2 | 0 | 0
  Any Swelling, D2 [N=118,117,111] | 15 | 9 | 24
  Grade 3 Swelling, D2 [N=118,117,111] | 0 | 0 | 0
  Any Pain, Across [N=119,119,116] | 91 | 95 | 98
  Grade 3 Pain, Across [N=119,119,116] | 7 | 6 | 12
  Any Redness, Across [N=119,119,116] | 48 | 50 | 53
  Grade 3 Redness, Across [N=119,119,116] | 2 | 0 | 1
  Any Swelling, Across [N=119,119,116] | 26 | 28 | 39
  Grade 3 Swelling, Across [N=119,119,116] | 0 | 0 | 0

5. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were Fatigue, Gastrointestinal (meaning nausea, vomiting, diarrhoea and/or abdominal pain), Headache, Myalgia, Shivering and Temperature (temperature higher than [≥] 37.5 degrees Celsius [°C]). "Any" = occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. "Related" = occurrence of the specified symptom assessed by the investigators as causally related to vaccination. "Grade 3 Fatigue" = fatigue that prevented normal activity. "Grade 3 Gastrointestinal" = gastrointestinal that prevented normal every day activities. "Grade 3 Headache" = headache that prevented normal activity. "Grade 3 Myalgia" = myalgia that prevented normal activity. "Grade 3 Shivering" = shivering that prevented normal activity. "Grade 3 Temperature" = temperature higher than (>) 39.0°C.
Time Frame: During the 7 day period (Days 0-6) following each dose (D)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects
  Any Fatigue, D1 [N=119,119,115] | 42 | 50 | 46
  Grade 3 Fatigue, D1 [N=119,119,115] | 3 | 1 | 0
  Related Fatigue, D1 [N=119,119,115] | 37 | 49 | 38
  Any Gastrointestinal, D1 [N=119,119,115] | 22 | 17 | 17
  Grade 3 Gastrointestinal, D1 [N=119,119,115] | 3 | 1 | 0
  Related Gastrointestinal, D1 [N=119,119,115] | 19 | 14 | 12
  Any Headache, D1 [N=119,119,115] | 35 | 39 | 34
  Grade 3 Headache, D1 [N=119,119,115] | 1 | 1 | 0
  Related Headache, D1 [N=119,119,115] | 31 | 31 | 26
  Any Myalgia, D1 [N=119,119,115] | 43 | 38 | 46
  Grade 3 Myalgia, D1 [N=119,119,115] | 2 | 2 | 0
  Related Myalgia, D1 [N=119,119,115] | 36 | 33 | 40
  Any Shivering, D1 [N=119,119,115] | 25 | 25 | 29
  Grade 3 Shivering, D1 [N=119,119,115] | 1 | 0 | 0
  Related Shivering, D1 [N=119,119,115] | 22 | 22 | 26
  Any Temperature, D1 [N=119,119,115] | 21 | 22 | 14
  Grade 3 Temperature, D1 [N=119,119,115] | 1 | 0 | 0
  Related Temperature, D1 [N=119,119,115] | 19 | 21 | 13
  Any Fatigue, D2 [N=118,117,111] | 43 | 46 | 59
  Grade 3 Fatigue, D2 [N=118,117,111] | 4 | 4 | 4
  Related Fatigue, D2 [N=118,117,111] | 41 | 41 | 56
  Any Gastrointestinal, D2 [N=118,117,111] | 14 | 5 | 12
  Grade 3 Gastrointestinal, D2 [N=118,117,111] | 0 | 1 | 1
  Related Gastrointestinal, D2 [N=118,117,111] | 14 | 5 | 10
  Any Headache, D2 [N=118,117,111] | 36 | 27 | 37
  Grade 3 Headache, D2 [N=118,117,111] | 2 | 3 | 5
  Related Headache, D2 [N=118,117,111] | 32 | 22 | 33
  Any Myalgia, D2 [N=118,117,111] | 48 | 42 | 43
  Grade 3 Myalgia, D2 [N=118,117,111] | 5 | 2 | 3
  Related Myalgia, D2 [N=118,117,111] | 46 | 39 | 38
  Any Shivering, D2 [N=118,117,111] | 25 | 23 | 35
  Grade 3 Shivering, D2 [N=118,117,111] | 3 | 3 | 3
  Related Shivering, D2 [N=118,117,111] | 24 | 20 | 31
  Any Temperature, D2 [N=118,117,111] | 20 | 16 | 26
  Grade 3 Temperature, D2 [N=118,117,111] | 0 | 0 | 2
  Related Temperature, D2 [N=118,117,111] | 19 | 16 | 24
  Any Fatigue, Across [N=119,119,116] | 54 | 63 | 71
  Grade 3 Fatigue, Across [N=119,119,116] | 7 | 5 | 4
  Related Fatigue, Across [N=119,119,116] | 49 | 57 | 65
  Any Gastrointestinal, Across [N=119,119,116] | 27 | 20 | 27
  Grade 3 Gastrointestinal, Across [N=119,119,116] | 3 | 2 | 1
  Related Gastrointestinal, Across [N=119,119,116] | 26 | 17 | 21
  Any Headache, Across [N=119,119,116] | 47 | 47 | 53
  Grade 3 Headache, Across [N=119,119,116] | 2 | 4 | 5
  Related Headache, Across [N=119,119,116] | 41 | 38 | 45
  Any Myalgia, Across [N=119,119,116] | 63 | 57 | 64
  Grade 3 Myalgia, Across [N=119,119,116] | 7 | 4 | 3
  Related Myalgia, Across [N=119,119,116] | 57 | 52 | 57
  Any Shivering, Across [N=119,119,116] | 37 | 35 | 48
  Grade 3 Shivering, Across [N=119,119,116] | 4 | 3 | 3
  Related Shivering, Across [N=119,119,116] | 34 | 29 | 43
  Any Temperature, Across [N=119,119,116] | 32 | 32 | 33
  Grade 3 Temperature, Across [N=119,119,116] | 1 | 0 | 2
  Related Temperature, Across [N=119,119,116] | 29 | 31 | 30

6. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 30 Days (Day 0-29) following vaccination
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects
  Any AEs | 27 | 27 | 23
  Grade 3 AEs | 4 | 4 | 4
  Related AEs | 9 | 5 | 7

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity.
Time Frame: From first vaccination up to one month (30 Days) post last vaccination
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects | 0 | 4 | 8

8. Secondary Outcome: Number of Subjects With SAE(s).
Description: as for outcome 7
Time Frame: Starting from 30 Days post last vaccine administration up to study end at Month 24
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects | 5 | 6 | 4

9. Secondary Outcome: Number of Days With Solicited Local Symptoms.
Description: Each dose was abbreviated as follows: D1 = Dose 1, D2 = Dose 2.
Time Frame: During the 7 Days (Day 0-6) following vaccination
Population: as for outcome 4
Measure: Number; unit: Days
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Days
  Days with Pain, D1 | 84 | 77 | 80
  Days with Pain, D2 | 71 | 83 | 87
  Days with Redness, D1 | 37 | 39 | 32
  Days with Redness, D2 | 28 | 27 | 37
  Days with Swelling, D1 | 17 | 23 | 25
  Days with Swelling, D2 | 15 | 9 | 24

10. Secondary Outcome: Number of Days With Solicited General Symptoms.
Description: Each dose was abbreviated as follows: D1 = Dose 1, D2 = Dose 2.
Time Frame: During the 7 Days (Day 0-6) following vaccination
Population: as for outcome 4
Measure: Number; unit: Days
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Days
  Days with Fatigue, D1 | 42 | 50 | 46
  Days with Fatigue, D2 | 43 | 46 | 59
  Days with Gastrointestinal, D1 | 22 | 17 | 17
  Days with Gastrointestinal, D2 | 14 | 5 | 12
  Days with Headache, D1 | 35 | 39 | 34
  Days with Headache, D2 | 36 | 27 | 37
  Days with Myalgia, D1 | 43 | 38 | 46
  Days with Myalgia, D2 | 48 | 42 | 43
  Days with Shivering, D1 | 25 | 25 | 29
  Days with Shivering, D2 | 25 | 23 | 35
  Days with Temperature, D1 | 21 | 22 | 14
  Days with Temperature, D2 | 20 | 16 | 26

11. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs).
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Dose 1 up to one month (30 days) following the last vaccine dose administration (Dose 2)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects With pIMDs.
Description: as for outcome 11
Time Frame: From one month (30 Days) following the last vaccine administration up to study end at Month 24
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Number analyzed (Participants) | 119 | 119 | 116
Subjects | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected during the entire study period (up to Month 24). Other Adverse Events were collected during the 30 Day post-vaccination period (Day 0 - Day 29).
Arm/Group | GSK1437173A-0,2 M Group | GSK1437173A-0,6 M Group | GSK1437173A-0,12 M Group
Serious Adverse Events (participants affected / at risk) | 5/119 | 9/119 | 12/116
Other Adverse Events (participants affected / at risk) | 107/119 | 106/119 | 107/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A-0,2 M Group (N=119) | GSK1437173A-0,6 M Group (N=119) | GSK1437173A-0,12 M Group (N=116)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A-0,2 M Group (N=119) | GSK1437173A-0,6 M Group (N=119) | GSK1437173A-0,12 M Group (N=116)
Chills (General disorders) | 37 (50) | 35 (48) | 48 (64)
Erythema (Skin and subcutaneous tissue disorders) | 48 (65) | 51 (69) | 53 (69)
Fatigue (General disorders) | 54 (85) | 63 (98) | 71 (105)
Gastrointestinal disorder (Gastrointestinal disorders) | 27 (36) | 20 (22) | 27 (29)
Headache (Nervous system disorders) | 48 (72) | 48 (68) | 53 (72)
Myalgia (Musculoskeletal and connective tissue disorders) | 63 (91) | 57 (80) | 64 (89)
Pain (General disorders) | 91 (155) | 95 (161) | 98 (167)
Pyrexia (General disorders) | 32 (41) | 32 (38) | 33 (40)
Swelling (General disorders) | 26 (32) | 28 (33) | 39 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.